CLINICAL TRIAL: NCT01397708
Title: A Phase I/II, Open Label Study of Ad-RTS-hIL-12, an Adenovirus Vector Engineered to Express hIL-12, in Combination With an Oral Activator Ligand, in Subjects With Unresectable Stage III or IV Melanoma
Brief Title: Safety Study of Adenovirus Vector Engineered to Express hIL-12 in Combination With Activator Ligand to Treat Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADA1001; ATI001-101 (Other: ZIOPHARM)
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Melanoma
Keywords: Melanoma; Unresectable
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INXN-1001 in combination with INXN-2001 (Experimental): Intratumoral injections of INXN-2001 (Ad-RTS-hIL-12) at a constant dose in combination with inter-cohort escalating doses of INXN-1001 (activator ligand).
  Interventions: Biological: INXN-2001; Drug: INXN-1001

INTERVENTIONS:
Biological: INXN-2001 — * approximately 1.0 x 1012 viral particles (vp) per injection
  * one intratumoral injection of INXN-2001 per study cycle
  * maximum of 6 study cycles
  Other Names: Ad-RTS-hIL-12
Drug: INXN-1001 — * 4 dose cohorts (5mg/day, 20mg/day, 100mg/day, and 160mg/day)
  * 7 oral daily doses of INXN-1001 per study cycle
  * maximum of 6 study cycles
  * 1 Expansion cohort at a single dose level at or below MTD (160mg/day)
  Other Names: Activator Ligand

SUMMARY:
This research study involves two investigational drugs, an Activator Ligand (INXN-1001) in combination with an Adenovirus Vector Engineered to Express hIL-12 (INXN-2001). IL-12 is a protein that may improve the body's natural response to disease by enhancing the ability of the immune system to kill tumor cells and may interfere with blood flow to the tumor.

The main purpose of this study is to evaluate the safety and tolerability of tumor injections of INXN-2001 given in combination with different doses of INXN-1001.

DETAILED DESCRIPTION:
Single-arm, open label, Phase I/II dose escalation study of intratumoral injections INXN-2001 and oral INXN-1001 in subjects with unresectable Stage III or IV melanoma.

Four sequential dose escalation cohorts of INXN-1001 in combination with a fixed dose of INXN-2001 are planned. Subject enrollment and dose escalation will proceed according to a standard 3+3 design.

Approximately 15 additional subjects will be enrolled as an expansion cohort at a single dose level at or below the MTD.

* Safety and tolerability will be assessed by the incidence and severity of adverse events.
* The antitumor activity of study treatment will be assessed according to RECIST v1.1 guidelines. Additional assessment of anti-tumor activity will be explored based on total measurable tumor burden.
* Immunological and biological markers of response will include examinations of tumor biopsy samples, cytokine levels, peripheral blood mononuclear cells (PBMC) and antibody response to INXN-2001.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of all races ≥ 18 years of age, who have provided written informed consent prior to completing any study specific procedure.
* Unresectable Stage III or Stage IV melanoma arising from any site other than ocular melanoma.
* A minimum of 2 accessible nonvisceral lesions (shortest diameter ≥1 cm) or palpable tumor-involved lymph nodes (shortest diameter ≥1.5 cm).
* ECOG performance status of 0 or 1 (Appendix 1).
* Adequate bone marrow, liver, and renal function.
* An expected survival of at least approximately 6 months.
* Male and female subjects must agree to use a highly reliable method of birth control (expected failure rate less than 5% per year) from the screening visit through 28 days after the last dose of study drug.

Exclusion Criteria:

* Any prior anti-cancer therapy or investigational agent within 28 days prior to the first dose of study drug. (NOTE: For the expansion cohort ONLY, if subjects received ipilimumab, a 90-day washout period since last dose of ipilimumab is required. If subjects received other immunomodulating therapies (eg, anti-PD1 antibodies), the medical monitor should be contacted and an evaluation will be made.)
* Clinically significant infection requiring systemic antibacterial, antifungal, or antiviral therapy within 2 weeks of the first dose of study drug.
* History of HIV infection.
* Active autoimmune disease requiring steroids (>10 mg prednisone or comparable) or other immunosuppressive therapy (e.g., methotrexate, etc.).
* Documented symptomatic brain metastases. Screening for brain lesions by CT or MRI is not required for all potential subjects; however, if there are any neurological signs or symptoms consistent with brain metastases, then a brain CT or MRI should be performed as clinically indicated.
* Any medications that induce, inhibit or are substrates of CYP450 3A4 within 7 days prior to the first dose of study drug.
* Prior history of hematopoietic stem cell transplant or organ allograft.
* Other concurrent clinically active malignant disease, with the exception of other cancers of the skin.
* Females who are nursing or pregnant.
* Subjects who have a history of hypersensitivity that may relate to any component of the study drugs, e.g. to benzoic acid since INXN-1001 contains two benzene rings.
* Unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a subject and/or their compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaymes Holland, Study Director — Alaunos Therapeutics
Locations (9):
- United States (9):
  - The Angeles Clinic, Los Angeles, California
  - Oncology Specialists, Park Ridge, Illinois
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Washington University, St Louis, Missouri
  - Atlantic Melanoma Center, Morristown, New Jersey
  - St. Lukes, Easton, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Fletcher Allen Health, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: 5mg QD: Phase I (Dose escalation): Ad-RTS-hIL-12 + Veledimex 5 mg QD for 7 days every 21 days
- Phase 1: 20mg QD: Phase I (Dose escalation): Ad-RTS-hIL-12 + Veledimex 20 mg QD for 7 days every 21 days
- Phase 1: 100mg QD: Phase I (Dose escalation): Ad-RTS-hIL-12 + Veledimex 100 mg QD for 7 days every 21 days
- Phase 1: 160mg QD: Phase I (Dose escalation): Ad-RTS-hIL-12 + Veledimex 160mg QD for 7 days every 21 days
- Phase II Group 1: 160mg QD: Phase II (Group 1): Ad-RTS-hIL-12 + Veledimex 160mg QD for 7 days every 21 days
- Phase II Group 2: 160mg QOD: Phase II (Group 2): Ad-RTS-hIL-12 + Veledimex 160mg QOD for 14 days every 28 days
- Phase II Group 2: 120mg QOD: Phase II (Group 2): Ad-RTS-hIL-12 + Veledimex 120mg QOD for 14 days every 28 days
- Phase II Group 2: 80mg QOD: Phase II (Group 2): Ad-RTS-hIL-12 + Veledimex 80mg QOD for 14 days every 28 days
Period: Overall Study
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Started | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2
Completed | 3 | 3 | 1 | 3 | 3 | 4 | 2 | 1
Not Completed | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population is defined as all patients who receive at least one INXN-1001 capsule or, in the event an injection of INXN-2001 is administered before an INXN-1001 capsule is taken, at least one injection of INXN-2001.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2 | 26
Age, Continuous [Median (Full Range); unit: years] | 45.0 [33 to 69] | 71.0 [57 to 94] | 73.0 [71 to 79] | 59.5 [59 to 74] | 70.0 [22 to 90] | 54.0 [39 to 66] | 63.0 [45 to 74] | 55.0 [27 to 83] | 64.0 [22 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 1 | 0 | 2 | 0 | 0 | 8
  Male | 3 | 1 | 0 | 3 | 4 | 2 | 3 | 2 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 3 | 3 | 4 | 4 | 4 | 3 | 2 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 182.50 (12.471) | 172.27 (12.329) | 154.90 (3.439) | 170.65 (12.619) | 174.95 (11.103) | 171.10 (10.370) | 174.00 (8.900) | 186.10 (5.515) | 172.69 (12.080)
Weight [Mean (Standard Deviation); unit: kg] | 88.30 (15.679) | 77.27 (21.388) | 59.60 (8.931) | 87.65 (11.577) | 80.53 (8.034) | 77.75 (20.012) | 81.03 (14.380) | 64.90 (1.556) | 78.16 (15.340)
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.408 (2.8240) | 25.645 (3.7322) | 24.796 (3.0863) | 30.542 (6.4765) | 26.508 (3.7585) | 26.541 (6.3030) | 26.660 (3.4900) | 18.777 (1.5615) | 26.248 (4.7793)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Evaluation will be based on the incidence, intensity, and type of Adverse Events (AEs). Clinically significant changes in the subjects' physical examinations, vital signs, and ECG evaluations, and clinical manifestations relevant to abnormal laboratory values will be captured as AEs.
Time Frame: From the signing of informed consent until 28 days after the last dose of study treatment, up to 28 weeks
Population: All safety analyses will be conducted on the Safety population. The Safety population is defined as all patients who receive at least one INXN-1001 capsule or, in the event an injection of INXN-2001 is administered before an INXN-1001 capsule is taken, at least one injection of INXN-2001.
  The Safety population will be used for the analysis of safety data based on the actual initial dose of INXN-1001 received.
Measure: Number; unit: participants
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2
participants
  Any TEAE | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2
  Drug-related TEAE | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2
  Drug-related Grade 3 or higher TEAE | 0 | 0 | 2 | 2 | 3 | 3 | 3 | 2
  TEAE leading to death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Treatment-emergent SAE | 0 | 0 | 1 | 2 | 3 | 3 | 2 | 2
  DLT | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0

2. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of INXN-1001 (Veledimex) in Cycle 1
Description: The area under the plasma concentration versus time curve from time 0 to the last measurable concentration (AUC0-t) for INXN-1001, calculated during the first treatment cycle.
Time Frame: Samples were collected in Cycle 1 on Day 1 (pre-dose and 0.5, 1, 2, 4, and 6 hours post-dose), Day 2 (pre-dose), Day 7 (pre-dose and 1-2 and 4-6 hours post-dose), and Day 8 (24 hours after the Day 7 dose).
Population: The PK Population includes all subjects who received at least one dose of INXN-1001 and had sufficient plasma concentration data to derive reliable PK parameters.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- 100 mg INXN-1001 (QD): Phase I (Dose escalation): Ad-RTS-hIL-12 + Veledimex 100 mg QD for 7 days every 21 days
- 160 mg INXN-1001 (QD): ATI001-101 (Melanoma): Ad-RTShIL-12 on Day 1 + INXN-1001 160 mg QDx7
- 160 mg INXN-1001 (QoD): ATI001-101 (Melanoma): Ad-RTShIL-12 on Day 1 + INXN-1001 160 mg QoDx7
- 120 mg INXN-1001 (QoD): ATI001-101 (Melanoma): Ad-RTShIL-12 on Day 1 + INXN-1001 20 mg QoDx7
- 80 mg INXN-1001 (QoD): ATI001-101 (Melanoma): Ad-RTShIL-12 on Day 1 + INXN-1001 80 mg QoDx7
Arm/Group | 100 mg INXN-1001 (QD) | 160 mg INXN-1001 (QD) | 160 mg INXN-1001 (QoD) | 120 mg INXN-1001 (QoD) | 80 mg INXN-1001 (QoD)
Number analyzed (Participants) | 3 | 8 | 4 | 3 | 2
ng*h/mL
  C1D1 AUC0-24 (ng*h/mL): number analyzed (Participants) | 2 | 6 | 4 | 3 | 2
  C1D1 AUC0-24 (ng*h/mL) | 11701 (2925) | 10225 (6214) | 16626 (12910) | 10322 (777) | 8364 (5771)
  C1D1 Dose-normalized m2/mg AUC0-24 (ng*h/mL): number analyzed (Participants) | 2 | 6 | 4 | 3 | 2
  C1D1 Dose-normalized m2/mg AUC0-24 (ng*h/mL) | 194 (16.1) | 148 (96) | 197 (105) | 193 (38) | 186 (135)
  C1D7 AUC0-t (ng*h/mL): number analyzed (Participants) | 3 | 3 | 3 | 1 | 2
  C1D7 AUC0-t (ng*h/mL) | 15900 (5960) | 14000 (1500) | 15700 (4640) | 11000 | 8945 (190)

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) was defined as the time in days from the first dose of study treatment to the first assessment of disease progression or death from any cause, whichever occurred first. Subjects who withdrew from the study were censored at the date of their last non-progressive disease assessment. The final analysis was performed using Kaplan-Meier methodology to determine the median PFS.
Time Frame: From the first dose of study treatment for up to 1 year.
Population: Subjects with at least one post baseline evaluation. Two subjects were enrolled in the 80 mg QOD arm. Both discontinued study treatment early and did not receive post-baseline tumor assessments. One subject completed scheduled visits but had no RECIST-evaluable imaging and was censored at baseline. Therefore, 0 subjects from this arm were included in the PFS analysis. The overall PFS-evaluable population included 17 subjects across all arms.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 3 | 1 | 0
Days | 79.0 [71.0 to 79.0] | 76.5 [74.0 to 79.0] | 29.5 [15.0 to 44.0] | 58.0 [57.0 to 64.0] | 64.0 [38.0 to 64.0] | 77.0 [27.0 to 162.0] | 91.0 [91.0 to 91.0] |

4. Secondary Outcome: Change From Baseline in Tumor IL-12 Messenger RNA (mRNA) Expression Change in IL-12 mRNA Expression Level (Arbitrary Units)
Description: Tumor biopsy samples were analyzed for IL-12 mRNA expression using quantitative real-time polymerase chain reaction (qRT-PCR).
  Expression levels were normalized to the housekeeping gene ACTB (β-actin) and quantified using the ΔΔCt method.
  For each participant, the median ΔΔCt-based fold-change from baseline to post-treatment was calculated.
  These individual participant-level medians were then averaged to derive the mean of medians (measure type) across all participants within each arm/group.
  The reported values therefore reflect the mean of medians in arbitrary units (AU), representing relative IL-12 mRNA expression normalized to ACTB- calculated as 2^(-ΔΔCt) fold-change relative to baseline
  Not all subjects in each arm contributed evaluable IL-12 mRNA expression data due to biopsy availability and RNA quality.
Time Frame: Baseline (Screening) and at the Post-Treatment Safety Assessment (approximately 28 days after the end of Cycle 1).
Population: The analysis was performed on participants in the Safety Population who had paired (baseline and post-treatment) tumor biopsy samples suitable for qRT-PCR.
  Paired samples were required for inclusion.
  The number of participants analyzed per arm/group is lower than the total enrolled population because of limited biopsy availability, insufficient RNA yield, or RNA quality issues.
Measure: Mean (Standard Deviation); unit: Arbitrary Units (AU)
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Number analyzed (Participants) | 3 | 3 | 2 | 4 | 0 | 0 | 0 | 0
Arbitrary Units (AU)
  IL-12 mRNA levels: C1D1-7: number analyzed (Participants) | 1 | 3 | 2 | 4 | 0 | 0 | 0 | 0
  IL-12 mRNA levels: C1D1-7 | 7916 | 6296 (5958) | 2216 (1012) | 4327 (2516) |  |  |  |
  IL-12 mRNA levels: C1D8-15: number analyzed (Participants) | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 0
  IL-12 mRNA levels: C1D8-15 |  | 1716 (2968) | 3 (3) | 0 (1) |  |  |  |
  IL-12 mRNA levels: C2D1-7: number analyzed (Participants) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
  IL-12 mRNA levels: C2D1-7 |  | 8866 (15309) |  | 15 |  |  |  |
  IL-12 mRNA levels: C2D8-15: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  IL-12 mRNA levels: C2D8-15 | 2178 |  |  | 1 |  |  |  |
  IL-12 mRNA levels: C3D1-7: number analyzed (Participants) | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0
  IL-12 mRNA levels: C3D1-7 | 2648 | 162946 (239470) |  | 33 (41) |  |  |  |
  IL-12 mRNA levels: C3D8-15: number analyzed (Participants) | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0
  IL-12 mRNA levels: C3D8-15 |  | 82716 (116949) |  | 68 (116) |  |  |  |

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of INXN-1001 (Veledimex) in Cycle 1
Description: The maximum observed plasma concentration (Cmax) of INXN-1001 following oral administration, as determined from plasma sample analysis during the first treatment cycle
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 100 mg INXN-1001 (QD) | 160 mg INXN-1001 (QD) | 160 mg INXN-1001 (QoD) | 120 mg INXN-1001 (QoD) | 80 mg INXN-1001 (QoD)
Number analyzed (Participants) | 3 | 8 | 4 | 3 | 2
ng/mL
  C1D1 Cmax (ng/mL): number analyzed (Participants) | 2 | 6 | 4 | 3 | 2
  C1D1 Cmax (ng/mL) | 962 (323) | 738 (417) | 1284 (855) | 809 (120) | 636 (465)
  C1D1 Dose-normalized m2/mg Cmax (ng/mL): number analyzed (Participants) | 2 | 6 | 4 | 3 | 2
  C1D1 Dose-normalized m2/mg Cmax (ng/mL) | 16.2 (2.7) | 10.6 (6.3) | 15.5 (6.9) | 16.3 (3.7) | 14 (11)
  C1D1 C24h (ng/mL): number analyzed (Participants) | 2 | 6 | 4 | 3 | 2
  C1D1 C24h (ng/mL) | 81.9 (79.3) | 106 (105) | 86.8 (80.0) | 66.6 (38.6) | 78 (14)
  C1D7 Cmax (ng/mL): number analyzed (Participants) | 0 | 8 | 4 | 0 | 0
  C1D7 Cmax (ng/mL) |  | 1400 (150) | 1570 (464) |  |
  C1D7 Dose-normalized m2/mg Cmax (ng/mL): number analyzed (Participants) | 0 | 8 | 4 | 0 | 0
  C1D7 Dose-normalized m2/mg Cmax (ng/mL) |  | 16.2 (1.7) | 17.2 (5.6) |  |

6. Secondary Outcome: Change From Baseline in Peripheral Blood Cytotoxic T-Lymphocytes (CTLs)
Description: The percentage of Cytotoxic T-Lymphocytes (CTLs) within the CD8+ T-cell population was measured from serum samples by flow cytometry to assess changes in immune cell populations.
Time Frame: Baseline (Screening) and at Cycle 2, Day 7
Population: A total of 5 of the 26 treated subjects were included in this CTL analysis. Inclusion was based on the availability of paired peripheral blood samples at baseline and Cycle 2, Day 7
Measure: Mean (Standard Deviation); unit: % cells
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2
% cells
  CD3+CD8+ Median %cells at Screening |  | 30.90 (0) |  |  |  |  |  | 25.40 (0)
  CD3+CD8+ Median %cells at C2D15 |  | 33.00 (0) |  |  |  |  |  | 28.60 (0)
  CD3+CD8+ Median %cells at post-treatment safety assessment |  | 28.75 (0) |  |  |  |  |  | 24.00 (0)

7. Secondary Outcome: Change From Baseline in Peripheral Blood Regulatory T-cells (Tregs)
Description: The percentage of Regulatory T-cells (Tregs) in peripheral blood lymphocytes was measured from serum samples by flow cytometry to assess changes in immune cell populations.
Time Frame: Baseline (Screening) and at Cycle 2, Day 7.
Population: A total of 5 of the 26 treated subjects were included in this final analysis of peripheral blood Regulatory T-cell levels. Inclusion required availability of paired serum samples from Baseline and Cycle 2, Day 7.
Measure: Mean (Standard Deviation); unit: %cells
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Number analyzed (Participants) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2
%cells
  CD3+CD4+ Median %cells at Screening |  | 45.00 (0) |  |  |  |  |  | 37.30 (0)
  CD3+CD4+ Median %cells at C2D15 |  | 34.45 (0) |  |  |  |  |  | 48.30 (0)
  CD3+CD4+ Median %cells at post-treatment safety assessment |  | 31.25 (0) |  |  |  |  |  | 24.00 (0)

8. Secondary Outcome: Change From Baseline in Tumor Interferon-gamma (IFN-γ) Messenger RNA (mRNA) Expression
Description: Tumor biopsy samples were analyzed for IFN-γ mRNA expression using quantitative real-time polymerase chain reaction (qRT-PCR). This measure reports the fold change in expression from baseline. Due to very low or undetectable baseline IFN-γ expression in many tumor biopsy samples, the fold change values calculated by qRT-PCR using the delta-delta Ct method may result in large numeric values. All values reported reflect fold change from baseline and were calculated per the qRT-PCR assay standard procedures
Time Frame: Baseline (Screening) and at the Post-Treatment Safety Assessment (28 days after the end of Cycle 1).
Population: The analysis was performed on subjects from the Safety Population who had paired (baseline and post-treatment) tumor biopsy samples available for interferon-gamma (IFN-γ) mRNA analysis. A total of 12 of the 26 treated subjects were included in this final analysis. The number of participants analyzed per cohort reflects those who contributed data at any post-baseline time point, even if data were not available at all scheduled intervals.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Number analyzed (Participants) | 1 | 3 | 2 | 4 | 0 | 1 | 1 | 0
fold change
  IFN-gamma mRNA levels: C1D1-7: number analyzed (Participants) | 1 | 3 | 2 | 4 | 0 | 0 | 0 | 0
  IFN-gamma mRNA levels: C1D1-7 | 11 (0) | 89 (132) | 242 (340) | 30 (43) |  |  |  |
  IFN-gamma mRNA levels: C1D8-15: number analyzed (Participants) | 0 | 3 | 2 | 3 | 0 | 0 | 0 | 0
  IFN-gamma mRNA levels: C1D8-15 |  | 195 (293) | 239 (247) | 0 (0) |  |  |  |
  IFN-gamma mRNA levels: C2D1-7: number analyzed (Participants) | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
  IFN-gamma mRNA levels: C2D1-7 |  | 392 (617) |  | 33 (0) |  |  |  |
  IFN-gamma mRNA levels: C2D8-15: number analyzed (Participants) | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  IFN-gamma mRNA levels: C2D8-15 | 1 (0) | 68 (96) | 2 (0) | 24 (0) |  |  |  |
  IFN-gamma mRNA levels: C3D1-7: number analyzed (Participants) | 1 | 3 | 0 | 3 | 0 | 0 | 0 | 0
  IFN-gamma mRNA levels: C3D1-7 | 42 (0) | 83 (110) |  | 15 (13) |  |  |  |
  IFN-gamma mRNA levels: C3D8-15: number analyzed (Participants) | 0 | 2 | 0 | 3 | 0 | 1 | 1 | 0
  IFN-gamma mRNA levels: C3D8-15 |  | 417 (487) |  | 1 (2) |  | 89 (0) | 4 (0) |

9. Secondary Outcome: Ad-RTS-hIL-12 Vector Copy Numbers in Tumor Biopsy Samples
Description: To evaluate the presence of the viral vector in the tumor, biopsy samples were assessed for vector copy numbers using a quantitative polymerase chain reaction (qPCR) assay. The results are reported as the number of vector copies per 100 nanograms (ng) of deoxyribonucleic acid (DNA).
Time Frame: Day 2 of Cycle 1, Day 2 of Cycle 2, and Day 2 of Cycle 3.
Population: The analysis was performed on subjects from the Safety Population who had a tumor biopsy sample available for analysis at any of the specified time points. The number of subjects with available data varies by cohort and time point, and the Overall Number of Participants Analyzed for each cohort reflects the unique number of subjects in that cohort who contributed data at any time point.
Measure: Mean (Standard Deviation); unit: Vector Copies per 100 ng DNA
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Number analyzed (Participants) | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Vector Copies per 100 ng DNA
  Day 2 Cycle 1: number analyzed (Participants) | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Day 2 Cycle 1 | 1100000 (1800000) | 14000000 (25000000) | 100000000 |  |  |  |  |
  Day 2 Cycle 2: number analyzed (Participants) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
  Day 2 Cycle 2 |  | 12000000 (16000000) | 140000000 | 3000000 |  |  |  |
  Day 2 Cycle 3: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Day 2 Cycle 3 |  | 100000 | 100000 | 4000000 |  |  |  |

10. Secondary Outcome: Best Overall Response (BOR) by RECIST 1.1 Criteria
Description: Best Overall Response (BOR) was a pre-specified secondary endpoint assessed according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. BOR is the best response recorded from the start of treatment until disease progression. Responses include Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD).
Time Frame: From the first dose of study treatment for up to 1 year.
Population: Analysis of BOR was performed on all subjects who received at least one dose of study drug and were evaluable for response. Of the 26 treated patients, 15 were evaluable for Best Overall Response per RECIST v1.1. Subjects were excluded if no post-baseline tumor imaging was available. The Phase I 160 mg QD and Phase II 120 mg QOD and 80 mg QOD cohorts had no evaluable subjects at the data cutoff due to early discontinuation or pending imaging. No data were imputed
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 3 | 3 | 0 | 0
Participants
  Complete Response (CR) | 0 | 0 | 0 |  | 0 | 0 |  |
  Partial Response (PR) | 0 | 1 | 0 |  | 1 | 0 |  |
  Stable Disease (SD): | 1 | 1 | 2 |  | 1 | 0 |  |
  Progressive Disease (PD) | 2 | 1 | 1 |  | 1 | 3 |  |

11. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of INXN-1001 (Veledimex) in Cycle 1
Description: The time to reach the maximum observed plasma concentration (Tmax) of INXN-1001 following oral administration during the first treatment cycle.
Time Frame: as for outcome 2
Population: The analysis was performed on the PK Population, which includes all subjects who received at least one dose of INXN-1001 and had sufficient plasma concentration data to derive reliable PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 2
hours
  Cycle 1, Day 1: number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 0 | 3 | 2
  Cycle 1, Day 1 | 4 [2 to 6] | 4 [2 to 6] | 4 [4 to 6] | 4 [2 to 6] | 3 [2 to 4] |  | 4 [4 to 6] | 5 [4 to 6]
  Cycle 1, Day 7 | 4 [1 to 4] | 1 [1 to 2] | 4 [1 to 4] | 1.5 [1 to 4] | 1.5 [1 to 4] | 1 [1 to 2] | 1 [1 to 4] | 1.5 [1 to 2]

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events were monitored from the signing of informed consent through 28 days after the last dose of study drug (up to 28 weeks). Deaths (all-cause mortality) were monitored for up to 1 year following first dose
Arm/Group | Phase I: 5mg QD | Phase 1: 20mg QD | Phase 1: 100mg QD | Phase 1: 160mg QD | Phase II Group 1: 160mg QD | Phase II Group 2: 160mg QOD | Phase II Group 2: 120mg QOD | Phase II Group 2: 80mg QOD
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 1/4 | 0/4 | 0/4 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 2/4 | 3/4 | 3/4 | 2/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 4/4 | 4/4 | 4/4 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 5mg QD (N=3) | Phase 1: 20mg QD (N=3) | Phase 1: 100mg QD (N=3) | Phase 1: 160mg QD (N=4) | Phase II Group 1: 160mg QD (N=4) | Phase II Group 2: 160mg QOD (N=4) | Phase II Group 2: 120mg QOD (N=3) | Phase II Group 2: 80mg QOD (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: 5mg QD (N=3) | Phase 1: 20mg QD (N=3) | Phase 1: 100mg QD (N=3) | Phase 1: 160mg QD (N=4) | Phase II Group 1: 160mg QD (N=4) | Phase II Group 2: 160mg QOD (N=4) | Phase II Group 2: 120mg QOD (N=3) | Phase II Group 2: 80mg QOD (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphatic obstruction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (4) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (3) | 4 (4) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Perianal erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (3) | 3 (3) | 3 (4) | 4 (8) | 3 (5) | 3 (3) | 2 (3) | 0 (0)
Pyrexia (Gastrointestinal disorders) | 2 (5) | 1 (1) | 3 (4) | 2 (16) | 4 (7) | 3 (5) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (4) | 0 (0) | 2 (4) | 3 (9) | 3 (4) | 3 (5) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 1 (3) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine colour abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin K decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Contusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (3) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2013-04-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT01397708/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT01397708/SAP_001.pdf